CLINICAL TRIAL: NCT00819000
Title: TOP MS is a Study of Multiple Sclerosis Disease Management in Collaboration With Specialty Pharmacies
Brief Title: Therapy Optimization in Multiple Sclerosis (MS)
Acronym: TOP MS
Status: Completed | Type: Observational
Sponsor: Teva Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Other Study IDs: PM032
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Sclerosis
Keywords: Specialty Pharmacy; Therapy Management; Medication Compliance; Medication Adherence; Medication Persistence; Health Outcomes
MeSH Terms: conditions — Multiple Sclerosis; Medication Adherence | interventions — Glatiramer Acetate; Injections, Subcutaneous; Interferon beta-1a; Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated MS Subjects: Subjects who are treated with Glatiramer Acetate or Interferon (IFN)-β and receive their therapy from one of the participating Specialty Pharmacies
  Interventions: Drug: Glatiramer Acetate, IFN-beta 1a (IM), IFN-beta 1a (Subcutaneous), and IFN-beta 1b

INTERVENTIONS:
Drug: Glatiramer Acetate, IFN-beta 1a (IM), IFN-beta 1a (Subcutaneous), and IFN-beta 1b — MS therapies (listed above) used according to prescribers' instructions.
  Other Names: Copaxone®; Avonex®; Rebif®; Betaseron®

SUMMARY:
The purpose of this study is to determine if higher compliance and adherence rates to drug therapy for MS result in better health outcomes than lower rates of therapy compliance and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older, with a diagnosis of MS.
* Being treated with Glatiramer Acetate (GA) or (IFN)-β
* Receiving therapy from a participating Specialty Pharmacy

Exclusion Criteria:

* Has any contraindication to GA or IFN-β therapy, including pregnancy, trying to become pregnant, or breast feeding during the study
* Has received an experimental drug in the last thirty (30) days other than Fampridine SR (4-aminopyridine or 4-AP)
* Unlikely to be able to participate for the full two years of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are treated with Glatiramer Acetate or Interferon (IFN)-β and receive their therapy from one of the participating Specialty Pharmacies
Sampling Method: Non-Probability Sample
Enrollment: 2878 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Relationship of therapy Medication Possession Ratio (MPR), to patient outcomes | 12 months and 24 months

SECONDARY OUTCOMES:
Relationship of therapy adherence, defined as the accumulation of time from initiation to discontinuation of therapy and measured by time, to patient outcomes | 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MerriKay Oleen-Burkey, PhD, Study Chair — Teva Neuroscience, Inc.; Howard Zwibel, MD, Study Director — Neurologic Center of South Florida
Locations (3):
- United States (3):
  - Teva Investigational Site, Swartz Creek, Michigan
  - Teva Investigational Site, Columbus, Ohio
  - Teva Investigational Site, Carnegie, Pennsylvania

REFERENCES:
- [Derived] Cohen BA, Coyle PK, Leist T, Oleen-Burkey MA, Schwartz M, Zwibel H. Therapy Optimization in Multiple Sclerosis: a cohort study of therapy adherence and risk of relapse. Mult Scler Relat Disord. 2015 Jan;4(1):75-82. doi: 10.1016/j.msard.2014.09.214. Epub 2014 Oct 7. PMID 25787057
- [Derived] Coyle PK, Cohen BA, Leist T, Markowitz C, Oleen-Burkey M, Schwartz M, Tullman MJ, Zwibel H. Therapy optimization in multiple sclerosis: a prospective observational study of therapy compliance and outcomes. BMC Neurol. 2014 Mar 13;14:49. doi: 10.1186/1471-2377-14-49. PMID 24624979